CLINICAL TRIAL: NCT07346794
Title: The Underlying Neural Mechanism of TMS in Improving the Imbalance of "Microbiota-brain-gut Axis" in Alzheimer 's Disease Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMS82460341
Record Dates: First submitted 2025-12-16; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer's Disease; rTMS Stimulation
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing treatment (Experimental)
  Interventions: Procedure: TMS
- No treatment (No Intervention): The sham DLPFC-rTMS group will receive stimulation via a single helmet equipped with a sham coil, which is designed to induce similar noise and scalp sensations under the same parameters as the active stimulation group.

INTERVENTIONS:
Procedure: TMS — For the repetitive transcranial magnetic stimulation (rTMS) intervention, the dorsolateral prefrontal cortex (DLPFC) is selected as the stimulation target, with a stimulation frequency of 10 Hz; the intervention consists of 20 stimulation trains per day, 5 days per week, using a coil with a diameter of 9 cm, at an intensity of 80% of the motor threshold (minimum single-pulse intensity: 50 μV); each stimulation train lasts for 10 seconds, with an interval of 25 seconds between trains, and 20 trains per day totaling 2000 pulses. The treatment is administered once daily, five times a week, for 4 consecutive weeks, resulting in a total of 20 to 30 sessions, and the traditional "5-centimeter" method is adopted for localizing the DLPFC stimulation target.
  Arms: Patients undergoing treatment

SUMMARY:
What is this study about? This study focuses on Alzheimer's Disease (AD), a common neurodegenerative disease that affects memory, thinking, and daily life. We aim to explore whether a non-invasive treatment called Repetitive Transcranial Magnetic Stimulation (rTMS) can improve AD symptoms by regulating the "gut-brain-intestine axis" - a connection between gut bacteria, the brain, and the intestines.

Who can participate?

* **AD patients**: Aged 50-80, diagnosed with mild to moderate AD (MMSE score 18-27, MoCA score 10-26), with stable condition for at least 6 months, and able to cooperate with tests and treatment.
* **Healthy controls**: Aged 50-80, with normal cognitive function (MMSE ≥28, MoCA ≥27), no AD family history, and matched in age and gender with AD patients.

Those with epilepsy, severe mental illness, recent use of antibiotics/probiotics, or inability to complete MRI scans are not eligible.

What will participants experience?

* **AD patients**: Will be randomly divided into two groups. Both groups will receive 4 weeks of treatment (5 days/week) with a helmet-like device. One group gets real rTMS (safe magnetic stimulation to the brain), and the other gets sham stimulation (no effective magnetic field, but same sound/feel).
* **Healthy controls**: No treatment, but will complete the same tests as AD patients.
* **Tests during the study**: Cognitive assessments (memory, thinking skills via questionnaires), stool/blood sample collection (to check gut bacteria and body markers), and MRI scans (to look at brain structure/function) at baseline, 1 month, 3 months, 6 months, and 1 year.

What are the potential benefits?

* Free rTMS treatment (for AD patients), free MRI scans (valued at 700 RMB), and a 200 RMB subsidy.
* Free health checks (gut bacteria analysis, metabolic tests) and cognitive evaluations to understand personal health status.
* Contribution to developing new AD treatments that may help future patients.

Is it safe? rTMS is a clinically proven safe technique. Possible mild side effects (headache, scalp irritation) usually go away on their own. Sample collection (stool/blood) and MRI scans are non-invasive or minimally invasive. A professional team will monitor participants throughout to handle any issues.

For healthcare providers This is a multicenter, randomized, double-blind sham-controlled study (200 AD patients, 200 healthy controls). The primary goal is to explore rTMS's mechanism via the gut-brain-intestine axis, with MoCA score changes (6 months post-treatment) as the main outcome. It integrates multi-omics and neuroimaging data to provide evidence for AD's non-drug treatment.

ELIGIBILITY:
Inclusion Criteria:

* Dementia Patients: Conformed to internationally recognized diagnostic criteria for dementia (e.g., DSM-5, NINCDS-ADRDA)
* Diagnosed through clinical evaluation, neuropsychological scale assessments, and relevant examinations
* Aged ≥50 years and residing in Nanchang, Jiangxi
* With dementia-negative family history, no severe psychiatric or neurological disorders
* No history of major systemic diseases.

Exclusion Criteria:

* Unable to cooperate with all required examinations, intervention procedures, and sample collection during the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
MoCA score | Pre-intervention, Periprocedural, and Post-intervention at 1/3/6/12 months

IPD SHARING:
Plan to Share IPD: No